CLINICAL TRIAL: NCT05567510
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Metabolism and Excretion of [14C] BMS-986369 in Healthy Male Participants
Brief Title: A Study to Evaluate the Metabolism and Excretion of BMS-986369 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA073-002
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Healthy Participants
Keywords: BMS-986369; Drug absorption, distribution, metabolism, and excretion (ADME)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986369 (Experimental)
  Interventions: Drug: BMS-986369

INTERVENTIONS:
Drug: BMS-986369 — Specified dose on specified days

SUMMARY:
The purpose of the study is to assess mass balance, biotransformation, and excretion of BMS-986369 following study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants, of any race, determined by the investigator to have no significant deviation from normal in medical history or physical examination, which correspond to a condition that could potentially increase the risk for the participants, or jeopardize the integrity of the study data in 12-lead ECG measurements, vital signs, and clinical laboratory determinations at screening and/or check-in.
* Body mass index (BMI) of 18.0 through 33.0 kilogram meter squared (kg/m^2), inclusive. BMI = weight kg/height m^2.
* Absolute neutrophil counts must be greater than 2,500 per microliter (μL) at screening and Day -1.

Exclusion Criteria:

* Any significant acute or chronic medical illness that presents a potential risk to the participant in the opinion of the investigator and/or may compromise the objectives of the study.
* Current or recent (within 3 months of study intervention administration) history of clinically significant endocrine, GI, cardiovascular, peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities/diseases.
* Participant has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion (ADME) (eg, bariatric procedure). Appendectomy, cholecystectomy, and uncomplicated hernia repair are acceptable. Prior procedures of unclear ADME significance should be reviewed with the Sponsor's Medical Monitor.

Prior/Concomitant Therapy

* Participant has participated in another investigational trial within 4 weeks prior to screening. For participants who have participated in an investigational trial where no trial drug was administered or invasive procedure performed, the waiting interval may be eliminated.
* Participant has received a vaccination, including coronavirus disease 2019 (COVID-19) vaccine, within 30 days prior to the IP dose or plans to receive vaccination within 2 months after dosing.
* Participant has used a prescribed systemic or topical medication (eg, analgesics, anesthetics, anti-coagulants, etc.) within 30 days prior to the first dose administration. Exceptions may be made on a case-by-case basis if considered not to interfere with study objectives as agreed to by the investigator and Sponsor's Medical Monitor.
* Use of CYP3A inducers (eg, St. John's wort) and inhibitors (eg, grapefruit juice) within 30 days prior to dosing.
* Participant has used any non-prescribed systemic or topical medications (for example, vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration. Exceptions may be made on a case-by-case basis if considered not to interfere with study objectives as agreed to by the investigator and Sponsor's Medical Monitor (eg, occasional use of acetaminophen).
* Participant has received immunization with a live or live-attenuated vaccine within 2 months prior to dosing or is planning to receive immunization with a live or non-live vaccine for 2 months following dosing.
* Participated in a radiolabeled drug study, where exposures are known to the investigator, within the previous 4 months prior to check-in (Day -1); or participated in a radiolabeled drug study, where exposures are not known to the investigator, within the previous 6 months prior to check-in (Day -1). The total 12-month exposure from this study and a maximum of 2 other previous studies within 4 to 12 months of this study will be within the CFR-recommended levels considered safe, per US Title 21 CFR 361.15: less than 5,000 mrem whole body annual exposure, with consideration given to the half-lives of the previous radiolabeled study drugs received.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Total radioactivity recovered in whole blood | Up to 22 days
Total radioactivity recovered in plasma | Up to 22 days
Total radioactivity recovered in urine | Up to 22 days
Total radioactivity recovered in feces | Up to 22 days
Total radioactivity recovered in vomit | Up to 22 days
Maximum observed plasma concentration (Cmax) | Up to 22 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to 22 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 22 days
Total radioactivity recovered in whole blood to plasma ratio | Up to 22 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 28 days
Number of participants with serious adverse events (SAEs) | Up to 28 days
Number of participants with vital sign abnormalities | Up to 28 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 28 days
Number of participants with clinical laboratory test abnormalities | Up to 28 days
Number of participants with physical examination abnormalities | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Labcorp Clinical Research Unit - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm